CLINICAL TRIAL: NCT01019213
Title: Acute and Chronic Effect of His-pacing in Consecutive Patients With AV-block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Mads Brix Kronborg, Dr., Aarhus University Hospital Skejby
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07-4-B695-A1464-22378
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Atrioventricular Block
Keywords: His-pacing
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Septal pacing (Placebo Comparator): Septal lead will be activated.
  Interventions: Other: Septal pacing
- His-pacing (Experimental): His lead will be activated 80 ms before septal lead
  Interventions: Other: His lead activated

INTERVENTIONS:
Other: Septal pacing — Septal lead activated
  Other Names: Septal lead
  Arms: Septal pacing
Other: His lead activated — His lead will be activated 80 ms before septal lead
  Other Names: His lead
  Arms: His-pacing

SUMMARY:
Conventional right ventricular (RV) apical pacing may result in asynchronous ventricular contraction with delayed left ventricular activation, interventricular motion abnormalities, and worsening of left ventricular ejection fraction. His pacing is preserving a synchronous contraction and may prevent a decrease in left ventricular ejection fraction.

Hypothesis: His-pacing preserves left ventricular function and is a feasable alternative compared to RV septal septal pacing in patients with AV-block.

DETAILED DESCRIPTION:
Conventional right ventricular apical pacing may result in asynchronous ventricular contraction with delayed left ventricular activation, interventricular motion abnormalities, and worsening of left ventricular ejection fraction. His pacing is preserving a synchronous contraction and may prevent a decrease in left ventricular ejection fraction.

The aims of our crossover, double-blinded, randomized study is to evaluate the feasibility and long-term safety of permanent His pacing and to compare the effects on left ventricular ejection fraction of permanent His pacing with those of conventional right septal stimulation after 12 months treatment in patients with 2nd or 3rd degree AV-block.

ELIGIBILITY:
Inclusion Criteria:

* 2nd or 3rd degree Av block

Exclusion Criteria:

* QRS > or = 120 ms
* Indication for cardiac resynchronization therapy (CRT) or implantable cardioverter defibrillator (ICD)
* chronic atrial fibrillation
* Pregnant
* Expected heart surgery < 2 years
* Expected survival > 2 years
* Patients that have been His ablated
* Serious comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 12 months

SECONDARY OUTCOMES:
Quality of life | 12 months
Synchrony by echocardiography | 12 months
New York Heart Association (NYHA) class | 12
6-minute hall walk test | 12

CONTACTS AND LOCATIONS:
Overall Officials: Torsten T Nielsen, Professor, Study Chair — Dept. B Skejby Hospital; Jens C Nielsen, Phycisian, Study Chair — Aarhus university Hospital Skajby; Mads B Kronborg, Phycisian, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Dept. of cardiology Skejby Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Kronborg MB, Mortensen PT, Poulsen SH, Gerdes JC, Jensen HK, Nielsen JC. His or para-His pacing preserves left ventricular function in atrioventricular block: a double-blind, randomized, crossover study. Europace. 2014 Aug;16(8):1189-96. doi: 10.1093/europace/euu011. Epub 2014 Feb 7. PMID 24509688